CLINICAL TRIAL: NCT00422552
Title: An Exploratory, Double-Blind Comparison of Inspiratory Capacity (IC) and FEV1 in COPD Patients Following Single Dose Administration of Indacaterol and Placebo and Open Label b.i.d. Administration of Formoterol
Brief Title: Effect of Indacaterol on Inspiratory Capacity and Lung Function in Patients With COPD Versus Placebo and Formoterol
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQAB149B2211
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: COPD
Keywords: inspiratory capacity, FEV1, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

INTERVENTIONS:
Drug: Indacaterol (QAB149)

SUMMARY:
The purpose of this study is to assess the change in inspiratory capacity and lung function in patients with chronic obstructive pulmonary disease when treated with indacaterol compared to placebo and formoterol.

ELIGIBILITY:
Inclusion Criteria:

* Male and post-menopausal female adults aged 40-80 years inclusive.
* Patients with a clinical diagnosis of COPD according to the Global Initiative for Chronic Lung Disease (GOLD) Guidelines (2005)
* Smoking history of at least 10 pack years (either smokers or ex-smokers).
* Able to perform reproducible spirometry maneuvers.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent.

Exclusion Criteria:

* COPD exacerbations within 6 weeks prior to dosing
* Concomitant lung disease such as asthma, requirement for long term oxygen treatment or history of lung reduction surgery.
* Medical conditions that would interfere with the performance of spirometry or may pose a potential hazard from performing spirometry.
* Any other medical condition that in the opinion of the Investigator may cause the patient to be unsuitable for completion of the study or place the patient at potential risk from being in the study, e.g. uncontrolled hypertension, unstable ischemic heart disease.
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-09

PRIMARY OUTCOMES:
Change from baseline in IC and percent predicted FEV1 at various timepoints over 24 hours

SECONDARY OUTCOMES:
Percent predicted FEV1 time course change over 24 hours
Mean maximal change in IC time course change over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Novartis Investigative site, Horsham, United Kingdom